CLINICAL TRIAL: NCT01170195
Title: Effectiveness of Licorice Extract Dietary Supplement on the Treatment of Postmenopausal Symptoms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: F&C Licorice Ltd (Other)
Responsible Party: Nir Kedem, F&C Licorice Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5459
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Postmenopausal Symptoms; Vaginal Dryness
Keywords: Postmenopausal; licorice; vaginal complaints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Calmera-Licorice Root Extract (Licogen) — 100 mg per day
  Other Names: Licogen

SUMMARY:
The purpose of the proposed study is to test the effect of Licorice Root Extract- Licogen on postmenopausal symptoms in postmenopausal women. Specifically, the study will also test the effect of the licorice extract on vaginal dryness.

DETAILED DESCRIPTION:
The estrogenic properties of glabridin, the major isoflavan in licorice root, were tested in view of the resemblance of its structure and lipophilicity to those of estradiol. The results indicate that glabridin is a phytoestrogen, binding to the human estrogen receptor and stimulating creatine kinase activity in rat uterus, epiphyseal cartilage, diaphyseal bone, aorta, and left ventricle of the heart. The stimulatory effects of 2.5-25 mg/animal glabridin were similar to those of 5 mg/animal estradiol. Chemical modification of glabridin showed that the position of the hydroxyl groups has a significant role in binding to the human estrogen receptor and in proliferation-inducing activity. Glabridin was found to be three to four times more active than 2*-O-methylglabridin and 4*-O-methylglabridin, and both derivatives were more active than 2*,4*- O-methylglabridin. The effect of increasing concentrations of glabridin on the growth of breast tumor cells was biphasic. Glabridin showed an estrogen receptor-dependent, growth-promoting effect at low concentrations (10 nM-10 mM) and estrogen receptor-independent antiproliferative activity at concentrations of >15 mM. This is the first study to indicate that isoflavans have estrogen-like activities. Glabridin and its derivatives exhibited varying degrees of estrogen receptor agonism in different tests and demonstrated growth-inhibitory actions on breast cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages 45-60,
2. Who are post-menopausal (proved by a laboratory test of FSH > 30 International units),
3. Patients who report having post-menopausal symptoms, who report having, at least 5-7 hot flushes per day, as well as wakeful night episodes and nocturnal sweating (measured by Greenscale or Cooperman Index).

Exclusion Criteria:

1. Female patients who are outside the age boundaries of 45-60,
2. Have FSH <30
3. Patients who presently have cancer of any kind,
4. Patients that are on any other treatment for relieving post-menopausal symptoms
5. Patients who have contraindication to Licorice.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
A beneficial effect of the licorice extract on postmenopausal symptoms (vasomotor symptoms, and nocturnal episodes) in symptomatic postmenopausal women | 20 weeks
  This outcome will be measured by:
  a diary in which she should report daily. The reporting would be for 3 parameters: number of hot flushes per day, wakefull night episodes and nocturnal sweating measured by Greens Climateric Scale
A beneficial effect of the licorice extract on vaginal complaints in symptomatic postmenopausal women | 20 weeks
  this objective will be measured by Pap Smear, Vaginal Ultra sound and vaginal PH

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kaplan, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel